CLINICAL TRIAL: NCT06096155
Title: Ambispective Study to Assess the Safety and the Performance of SAGITTA EVL R Stem
Acronym: 2022-09
Status: Recruiting | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-09_Sagitta EVL-R
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Hip Arthropathy
Keywords: Total Hip Prosthesis Revision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This clinical study is conducted to collect data on hip arthroplasty with the SAGITTA EVL-R revision femoral stems manufactured by SERF.

This study will confirm the performance and safety of the SAGITTA EVL R revision femoral stems within the framework of MDR 2017/745 and in relation to the recommendations of the MEDDEV guide 2.7.1. Rev 4 (Clinical Evaluation Guide), which provides for a systematic procedure to monitor clinical data in order to verify the claimed performance of medical devices.

The primary objective is to evaluate the long-term survival rate (7 to 10 years post-op +/- 2 years) of SAGITTA EVL R stems.

Secondary objectives are to :

* study long term patient satisfaction with their hip prosthesis,
* confirm the long-term safety of these implants by studying the possible complications observed,
* evaluate the performance of these implants using clinical scores.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old at the time of surgery,
* Patient implanted with a SAGITTA EVL R revision femoral stem within its indications between 01/01/2010 and 31/12/2015,
* Affiliated to French health insurance system

Exclusion Criteria:

* Patient who has rejected to the use of his/her personal data,
* Patient unable to understand the surgeon's instructions or to carry out the post-operative follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects who needed a revision of total hip arthroplasty, implanted with a SAGITTA EVL-R revision femoral stem according to instructions for use, over a period of time between 31/01/2010 and 31/12/2015.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate at mid/long term follow-up | At 7/10 years after surgery
  Assess the survival rate at 7/10 year-follow-up, whatever the cause of revision

SECONDARY OUTCOMES:
Patient's satisfaction | At 7/10 years after surgery
  Assessed by the surgeon through questionary with a 5 item-scale : very satisfied / satisfied / neither satisfied - nor unsatisfied / unsatisfied / very unsatisfied
Adverse events | At 7/10 years after surgery
  List type and occurence of adverse events
Oblivion of prosthesis | At 7/10 years after surgery
  Assess the degree of forgetfulness of the prosthesis using FJS-score : FJS stands for Forgotten Joint Score. The Forgotten Joint Score assessment consists of 12 questions and is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities
Pain release | At 7/10 years after surgery
  Evaluate pain using Modified Harris Hip Score :
  The global Harris Hip Score consists of a 0 to 100 points scale (100 points is the better outcome).
  The pain evaluation is picked out from the global Harris Hip Score. The pain item is scored on a 0 to 44 points scale (44 points means no pain).
Functional improvement | At 7/10 years after surgery
  Evaluate walking, limping and activities of daily life using Modified Harris Hip Score :
  The global Harris Hip Score consists of a 0 to 100 points scale (100 points is the better outcome).
  The functional improvement is picked out from the global Harris Hip Score and can be measured with 3 subscores :
  The walking ablility is assessed by 2 items (support for walk and distance walked, each one is scored a 0 to 11 points scale (11 points is the better outcome).
  The limping is assessed by a 0 to 11 points scale (11 points is the better outcome).
  The activities of daily life are assessed by a 0 to 14 points scale (14 points is the better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Loire Vendée Océan, Challans, Vendée, France